CLINICAL TRIAL: NCT06438588
Title: Effect of Fasting Mimicking Diet (FMD) on Immune Related Adverse Events for Cancer Patients on Immune Checkpoint Inhibitors: The FMD-ICI Feasibility Pilot Study
Brief Title: Fasting Mimicking Diet for Reducing Immune Related Adverse Events for Cancer Patients on Immune Checkpoint Inhibitors, FMD-ICI Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-012936; NCI-2024-03515 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-012936 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Diet Therapy; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (FMD) (Experimental): Patients receive nutrition counseling with a nutritionist over 60 minutes, receive FMD over 4 days for 3 cycles of immunotherapy and educational guidelines for day 5 to transition to a regular diet. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Interview; Other: Nutritional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Dietary Intervention — Given FMD
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Educational Intervention — Receive educational guidelines
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
Other: Nutritional Assessment — Receive nutrition counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial assesses an effective and translatable care model to understand and reduce the adverse effects that cancer patients experience during their treatment therapies and thereby enhance their well-being and quality of life. Excessive immune activation can affect multiple organs with the most common adverse effects being skin rash, diarrhea, colitis, fatigue, hypothyroidism and anorexia. A restrictive calorie diet, mostly of fat and complex carbohydrates, will mimic fasting and increase resiliency to protect patients from the adverse effects of cancer treatments, by managing the adverse side effects of immune checkpoint inhibitors (ICI) treatments in select cancer patients. The fast mimicking diet (FMD) (Xentigen®) is a calorie restrictive, low-calorie, low-protein, high complex carbohydrate, high-fat diet. The FMD program is a plant-based diet program designed to attain fasting-like effects while providing both macro- and micronutrients to minimize the burden of fasting and adverse effects. The FMD consists of 100% ingredients which are generally regarded as safe (GRAS) and comprises mainly of vegetable-based soups and broths, energy bars, energy drinks, cracker snacks, herbal teas, and supplements. Following a FMD may reduce the adverse effects that some cancer patients experience while following immunotherapy treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the impact of immunotherapy + FMD/Xentigen® on immune related adverse events rates (irAEs) (including immune-mediated colitis).

II. Appraise the impact of immunotherapy + FMD/Xentigen® on the patient's physical function and quality of life.

III. Evaluate the impact of immunotherapy + FMD/Xentigen® on surrogate markers of inflammation (i.e., fecal calprotectin) as a predictive marker of immune-mediated colitis.

OUTLINE:

Patients receive nutrition counseling with a nutritionist over 60 minutes, receive FMD over 4 days for 3 cycles of immunotherapy and educational guidelines for day 5 to transition to a regular diet. Patients undergo blood sample collection throughout the study.

Upon completion of study intervention, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing immunotherapy regardless of prior immunotherapy history
* Age ≥ 18 years
* Body mass index (BMI) > 19
* Histological confirmation of advanced staged malignancies (stage 3 or 4) appropriate for the following types of immunotherapy: PD-1 Antibody (nivolumab, pembrolizumab), PD-L1 Antibody (atezolizumab, avelumab, durvalumab), CTLA-4 Antibody (ipilimumab) or any combination thereof

Exclusion Criteria:

* Age < 18 years
* Pregnant women
* Nursing mothers
* Persons of childbearing potential who are unwilling to employ adequate contraception
* Patients will be excluded if they are on insulin due to diabetes [diabetic patients will be asked to monitor their glucose levels with a continuous glucose monitoring (CGM) device], if they have allergies to any of the components in the FMD, if there is unacceptable deterioration of their nutritional status and cancer progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Symptom Measurement | Up to 6 months
  Symptoms will be measured using a modified version of the Memorial Symptom Assessment Scale. The modified version will contain specific items related to side effects of immune checkpoint inhibitors (ICIs) including twelve GI symptoms, skin changes, and fatigue. The scale includes 24 items for which the participant reports on whether a symptom (e.g., pain, lack of energy, shortness of breath) occurred during the previous week, as well as any distress it may have caused. Questions are answered on a 0-4 or 0-4 scale (e.g., 1=Rarely, 2=Occasionally, 3=Frequently, 4=Almost Constantly).
Incidence of adverse events | Up to 6 months
  Will grade the severity of symptoms using the CTCAE v3.0 scale. Will report descriptive analysis of rates and means. Patients will also be asked to report on any incidences of involuntary fasting due to their symptoms.
Physical function | Up to 6 months
  Physical function will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function, a 10-item measure of mobility and extremity function that was specifically developed for use in cancer, populations. Items are scored from 1-5 each with higher scores indicating better physical function.
Quality of life - FACT-G | Up to 6 months
  Quality of life will be measured using the seven item Functional Assessment of Cancer Therapy (FACT-G), an abbreviated version of the FACT-G. Each item is scored from 0 (not at all) to 4 (very much). Higher overall scores correspond with better quality of life.
Fecal calprotectin | At baseline, week 12 and week 24
  Fecal calprotectin will be measured by patients who develop diarrhea or the gastrointestinal side effects. Will be obtained as standard of care to assess for immune mediated colitis if CTCAE v3.0 score is greater than 1.

CONTACTS AND LOCATIONS:
Overall Officials: Francis A. Farraye, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials